CLINICAL TRIAL: NCT02446080
Title: The Drink Milk Consumption Benefits With Culture Probiotic in the Treatment of Constipation Women
Brief Title: Drink Milk Consumption Benefits With Culture Probiotic in the Treatment of Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Univates (Other)
Responsible Party: Principal Investigator, Thaís Rodrigues Moreira, Nutrition Course Professor, Centro Universitário Univates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CUUnivates
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Constipation
Keywords: Constipation; Probiotics; Women
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic Group (Experimental): Milk drink with probiotic culture (150 mL/daily) for 60 days.
  Interventions: Dietary Supplement: Milk drink with probiotic culture
- Control Group (Active Comparator): Milk drink (150 mL/daily) for 60 days.
  Interventions: Dietary Supplement: Milk drink

INTERVENTIONS:
Dietary Supplement: Milk drink with probiotic culture — The Probiotc group was asked to drink 150 ml per day of dairy drinks with probiotic culture
  Arms: Probiotic Group
Dietary Supplement: Milk drink — The control group was asked to drink 150 ml per day of dairy drinks.
  Arms: Control Group

SUMMARY:
Constipation is defined as a disorder characterized by persistent difficulty to evacuate or a feeling of incomplete evacuation and / or infrequent bowel movements. Many factors contribute to the onset of constipation, such as changes in dietary intake and fluid intake, decrease in consumption of products containing fiber, intake of drugs or laxatives, decreased intestinal motility and physical inactivity. The objective was to evaluate the effect of consumption of dairy products with probiotics on constipation. Randomized double-blind clinical trial in the city of Bom Retiro do Sul / RS, Brazil. They were recruited 60 female patients aged 20-50 years after application of the Rome III criteria (World Gastroenterology Organization, 2010) and Range Bristol (World Gastroenterology Organisation, 2010) were diagnosed with constipation. Patients were randomized into two groups, where one group will receive the milk drink with probiotics and the other group will receive a probiotic milk drink without (control group). The milk beverage consumption period shall be 60 days where each patient will consume 150 ml of milk drink a day, with breakfast or morning snack.

DETAILED DESCRIPTION:
Randomized double blind clinical trial conducted at the health center of the city of Bom Retiro do Sul / RS, Brazil, from December 2014 to March 2015. The study began after approval by the Ethics Committee of the Research Center University Univates (COEP), Lajeado. Brazil. They were recruited 60 female patients aged 20-50 years after application of the Rome III criteria (World Gastroenterology Organization, 2010) and Range Bristol (World Gastroenterology Organisation, 2010) were diagnosed with constipation. Patients were randomized into two groups, where one group will receive the milk drink with probiotics and the other group will receive a probiotic milk drink without (control group). The milk beverage consumption period shall be 60 days where each patient will consume 150 ml of milk drink a day, with breakfast or morning snack. The milk drink was provided in the homes of participants and the health center of the city of Bom Retiro do Sul once a week. At the beginning of treatment and at the end of treatment that will last 60 days, will be delivered to Bristol Scale and the criteria of Rome III, so as to verify the improvement or not of constipation. Patients who agree to participate in the study signed a consent form IC. Will be the orientation for the volunteers not to consume yogurt and other cultured milks with probiotics, will also be oriented to maintain the same diet and lifestyle when they were constipated, thus, check for improvement in constipation with the use of probiotics .

Inclusion criteria: Having a diagnosis of constipation; Be aged between 20 and 50 years; being female.

Data collection brings no risk or damage to entrant, but can cause discomfort and embarrassment to meet the criteria of Rome III and Bristol Scale and the time that will have to spend 10 to 15 minutes. Such issues will be mitigated by the fact that the interview be individualized and the participant have at their disposal a private room to answer the questionnaires, only with the presence of the academic.

Participants will not obtain any financial benefit, only the benefits of milk drink with probiotics and how much consumption adds to your health. It is also important to note that participation in the study will not result in expenses.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of constipation;
* Have aged between 20 and 50 years;
* Being female.

Exclusion Criteria:

* Patients with diabetes;
* Patients pregnant and lactating women;
* Patients with diarrhea, with previous gastrointestinal disorders;
* Current or recent consumption of antibiotics, anti-inflammatory drugs, laxatives or other drugs;
* Patients with diseases that alter bowel habits, such as food allergies and intolerances, ulcerative colitis, chron's disease and irritable bowel syndrome.
* Patients who have lactose intolerance or dislike of milk drink.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Improvement of symptoms of constipation | 60 days
  Improvement of symptoms of constipation by ROME III criteria and Bristol scale.

SECONDARY OUTCOMES:
Increased number of bowel movements | 60 days
  Increased number of bowel movements per week and is quoted by ROME III criteria.